CLINICAL TRIAL: NCT03940222
Title: Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Brief Title: Comparison Between Patching and Interactive Binocular Treatment (IBiTTM) in Amblyopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamideh Sabbaghi, PhD student, Teacher Assistant, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBMU.12345
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: The New Treatment in Amblyopia Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-BiT group (Experimental): Amblyopic patients will play I-BiT games without patching.
  Interventions: Device: Interactive Binocular Treatment
- Placebo group (Placebo Comparator): Amblyopic patients will patch their dominant eye and they will play placebo I-BiT games.
  Interventions: Procedure: Patching Therapy

INTERVENTIONS:
Device: Interactive Binocular Treatment — The specified system which stimulate the fovea of the amblyopic eye directly by detailed and movable objects, while the fixation of the non- amblyopic eye will be focused on fixed targets.
  Arms: I-BiT group
Procedure: Patching Therapy — Patching of the dominant eye with better best corrected visual acuity
  Arms: Placebo group

SUMMARY:
The purpose of this study is to investigate the effect of amblyopia therapy on cases who will receive Interactive Binocular Treatment (IBiTTM) without patching compared with those who will receive standard patching of the dominant eye with placebo IBiTTM.

In this randomized clinical trial, 40 unilateral amblyopic children (3 to 10 years old) will be studied. All unilateral functional amblyopic children with best corrected visual acuity (BCVA) worse than 0.30 LogMAR at least in one eye or a difference of two BCVA lines of Snellen between the two eyes will be included and randomly will divide into the case (n=19) and control (n=21) groups. Cases will play I-BiT™ games, while controls will have standard patch therapy and will play with placebo IBiTTM for one month. All subjects will be underwent comprehensive ophthalmic examinations at baseline and at one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Functional amblyopia with BCVA less than 20/30 (0.3 LogMAR) at least in one eye
* A difference of two BCVA lines of Snellen between the two eyes

Exclusion Criteria:

* A history of penalization one month prior to the study
* Bilateral amblyopia
* BCVA less than 20/200
* Eccentric fixation
* Nystagmus
* Ocular deviation more than 10 prism diopter (pd)
* Organic amblyopia
* Uncooperative children those with
* Mental and physical disability
* Systemic diseases

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hamideh Sabbaghi, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No